CLINICAL TRIAL: NCT06218628
Title: Phase I Study Accessing the Safety of Pacritinib in Combination With Talazoparib in Patients With Myeloproliferative Neoplasms Unresponsive to Frontline JAK2 (Janus Kinase 2) Inhibition
Brief Title: Pacritinib w/ Talazoparib in Pts w/ Myeloproliferative Neoplasms Unresponsive to JAK2 Inhibition
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-1048; HM-224 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Chronic Myelomonocytic Leukemia; Polycythemia Vera; Essential Thrombocytosis
Keywords: Talazoparib; Pacritinib; JAK2 Inhibition; Myeloproliferative Neoplasm
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Polycythemia Vera; Thrombocythemia, Essential; Myeloproliferative Disorders | interventions — talazoparib; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level -1 (Experimental): 0.25 mg (PO, QD) Talazoparib (Days 1-7) 200 mg (PO, BID) Pacritinib (Day 1-28, Lead in dosing of Pacritinib day -7 for the first cycle of treatment)
  Interventions: Drug: Talazoparib; Drug: pacritinib
- Dose Level 1 (Experimental): 0.25 mg (PO, QD) Talazoparib (Days 1-14) 200 mg (PO, BID) Pacritinib (Day 1-28, Lead in dosing of Pacritinib day -7 for the first cycle of treatment)
  Interventions: Drug: Talazoparib; Drug: pacritinib
- Dose Level 2 (Experimental): 0.5 mg (PO, QD) Talazoparib (Days 1-14) 200 mg (PO, BID) Pacritinib (Day 1-28, Lead in dosing of Pacritinib day -7 for the first cycle of treatment)
  Interventions: Drug: Talazoparib; Drug: pacritinib
- Dose Level 3 (Experimental): 0.75 mg (PO, QD) Talazoparib (Days 1-14) 200 mg (PO, BID) Pacritinib (Day 1-28, Lead in dosing of Pacritinib day -7 for the first cycle of treatment)
  Interventions: Drug: Talazoparib; Drug: pacritinib
- Dose Level 4 (Experimental): 1 mg (PO, QD) Talazoparib (Days 1-14) 200 mg (PO, BID) Pacritinib (Day 1-28, Lead in dosing of Pacritinib day -7 for the first cycle of treatment)
  Interventions: Drug: Talazoparib; Drug: pacritinib

INTERVENTIONS:
Drug: Talazoparib — pacritinib in combination with talazoparib
  Other Names: talzenna
Drug: pacritinib — pacritinib in combination with talazoparib
  Other Names: vonjo

SUMMARY:
This is a prospective phase I dose-escalation study, with the primary objective to access the MTD and find the RP2D of talazoparib, given in combination with standard of care dosing of pacritinib.

DETAILED DESCRIPTION:
This is a prospective phase I dose-escalation study, with the primary objective to access the MTD and find the RP2D of talazoparib, given in combination with standard of care dosing of pacritinib. Subjects must have a diagnosis of a myeloproliferative neoplasm and progressed or become intolerant to any JAK2 directed therapy. To be eligible for the therapy, patients are required to consent to a bone marrow biopsy at the beginning of study treatment. The treatment protocol involves initiating pacritinib on day -7 (lead-in phase, starting day -7 for cycle 1) with a standard of care dose of 200mg twice daily (BID). Subsequently, talazoparib will be given on day 1 of the treatment cycle. Cohort 1 will enroll patients at the starting dose of 0.25mg talazoparib for 14 days (dose level 1) and DLT (dose-limiting toxicity) rate will inform the subsequent dose levels (DLs).

Investigators plan to use a Bayesian Optimal Interval Design (BOIN) to determine the maximum tolerated dose (MTD) in patients with Ph-MPNs (Philadelphia chromosome negative myeloproliferative neoplasms) who have either not responded to or cannot tolerate ruxolitinib monotherapy. Subjects who are currently receiving JAK2-directed therapy will undergo a one-day washout period before starting the study treatment, as abrupt discontinuation of JAK2 inhibition can lead to side effects. This brief interval allows for the resolution of any lingering effects before initiating the new treatment. A bone marrow aspirate and or biopsy will be obtained to assess response to therapy at the end of each cycle of treatment (28 days), prior to beginning the next cycle as per physician discretion. Peripheral blood and bone marrow mononuclear cells will be checked for γ-H2AX (histone H2A family X) at set time points as a biomarker assay to assess for DNA damage in the same manner as the pre-clinical models published in our previous studies. Patients may remain on study drug unless they experience an unacceptable toxicity, fail to show a benefit, or they attain remission and it is felt by the investigator that they can proceed to an allogenic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed primary myelofibrosis (PMF), post-polycythemia vera-myelofibrosis (PPV-MF), post-essential thrombocythemia-myelofibrosis (PET-MF), chronic myelomonocytic leukemia, polycythemia vera, or essential thrombocytosis according to the 2008 World Health Organization criteria
* Subject has at least 2 symptoms with a score ≥ 3 or a total score of ≥ 12, as measured by the MFSAF(Myelofibrosis Symptom Assessment Form) v4.0
* Subject classified as intermediate-2 or high-risk MF, as defined by the Dynamic International Prognostic Scoring System Plus (DIPSS+70).
* Age > 18 years.
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Subject must have received prior treatment with a single JAK2 inhibitor 4.1.6 for at least 12 weeks with documented disease progression OR subject must have appearance of new splenomegaly that is palpable to at least 5 cm below the left costal margin (LCM) in subjects with no evidence of splenomegaly prior to the initiation of any first line JAK2 inhibitor
* Baseline QTc (corrected QT interval) <0.47 seconds (Bazett formula)
* Patients must have normal organ function as defined in protocol.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Subjects must not be experiencing toxicity due to prior therapy that has not resolved to ≤Grade 1 by study registration, with the exception of sensory neuropathy related to previous systemic therapy exposure, alopecia and fatigue.
* Patients that have transformed to Acute Myeloid Leukemia defined by >20% blasts count on peripheral blood smear or bone marrow biopsy evaluation
* Uncontrolled inter-current illness including, but not limited to, any other malignancy (with the exception of hormonal therapy for breast cancer/prostate cancer in remission >1 year and for non-hormonal therapies for other cancers in remission for >3 years), other ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with history of hemorrhagic stroke and evidence of uncontrolled bleeding as well as bleeding disorder
* Known HIV positive patients on combination antiretroviral therapy are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2029-08-22 (Estimated); Study Completion 2030-08-27 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 6 years
  To define the maximum tolerated dose (MTD) of talazoparib in combination with standard of care dosing of pacritinib in order to establish a recommended phase II dose (RP2D).

SECONDARY OUTCOMES:
Rate of grade 3 or higher toxicity | 6 years
  Rate of grade 3 or higher toxicities occurring with the combination of talazoparib and pacritinib in patients with MPNs that have failed to respond to one line of JAK2 directed therapy.
Response rate | 6 years
  Response rate defined by a 35% or greater spleen volume reduction (SVR) or a >25% reduction in total symptom score (TSS) at week 24 (per IWG-MTR (International Working Group for Myelofibrosis Research and Treatment) criteria).
Disease control rate | 6 years
  Disease control rate, defined by improvement in quality of life measures, spleen size, and hematological recovery
Progression free survival | 6 years
  Progression free survival, defined as the time of enrollment to disease progression
Overall survival | 6 years
  Overall survival, defined by time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Peter Abdelmessieh, DO, MSc, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No